CLINICAL TRIAL: NCT05237934
Title: Tissue Procurement and Natural History Study of Neuroendocrine Neoplasms (NENs) Including Adrenocortical Carcinoma (ACC)
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000491; 000491-C
Record Dates: First submitted 2022-02-05; First posted 2022-02-14 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11-06

CONDITIONS: Neuroendocrine Tumors; Carcinoma, Neuroendocrine
Keywords: Clinical Outcome; Advice in the Management of Cancer; Patterns of Disease Progression; Response or Lack of Response to Therapeutic Interventions; Natural History
MeSH Terms: conditions — Neuroendocrine Tumors; Carcinoma, Neuroendocrine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1: Participants with confirmed/suspected NENs including ACC

SUMMARY:
Background:

Neuroendocrine neoplasm (NENs)are rare cancers arising from the neuroendocrine cells and can affect almost any part of the body. They vary from low grade neuroendocrine tumors (NETs) to high grade neuroendocrine carcinomas (NECs). These tumors often occur in the gastrointestinal tract, pancreas, lungs, adrenal medulla (pheochromocytomas) or adrenal cortex (adrenocortical cancer) and other areas of the body mentioned below:

* Gastroenteropancreatic neuroendocrine tumors (GEP-NET): stomach, duodenum, pancreas, colon, appendix, etc.
* Liver and gallbladder
* Adrenal tumors
* Pituitary gland
* Thyroid gland: medullary thyroid carcinoma
* Parathyroid tumors
* Pulmonary neuroendocrine tumors: typical and atypical carcinoid, small cell lung cancer (SCLC), large cell neuroendocrine carcinoma (LCNEC)
* Extrapulmonary small cell cancer
* Peripheral nervous system tumors: paraganglioma, neuroblastoma)
* Breast and genitourinary tract

Their rates are rising in the United States and worldwide. Researchers want to learn more about NENs through this natural history study.

Objective:

To study the natural history of people with NENs and obtain samples from them to learn more about the disease. The clinical management of all NETs is not standardized, with only a few FDA-approved therapies and we would like to learn which combination therapeutic approach should be used, how long treatment should be continued, and in what subgroup of NENs a particular treatment option should be used.

Eligibility:

People aged 18 and older who have or are suspected to have NENs or ACC.

Design:

Participants will be screened with a medical history.

Participants will have a physical exam. Their symptoms and their ability to perform their normal activities will be reviewed. They will have blood and urine tests.

Participants will receive recommendations for managing their disease and potential treatment options. They will be able to ask as many questions as they would like.

Participants may provide saliva and blood, a for research. They will give tumor samples from a previous surgery or biopsy.

Participants may have optional biopsies. During biopsies, cancer tissue will be obtained using a needle and syringe. Tissue will be taken from the liver, lung, or a lymph node. Participants may have an imaging scan or ultrasound to help locate the tumor or area to be biopsied. They will receive local anesthesia and may be sedated.

Participants will complete a questionnaire about their family medical history.

Participants will have follow-up visits every 12 months. They will have physical exams and give samples. If their health changes, they may have extra visits. If they cannot visit NIH, they (or their doctor) will be contacted by phone or email.

Participants will take part in the study for all their life.

DETAILED DESCRIPTION:
Background:

* Neuroendocrine neoplasms (NENs) are divided into neuroendocrine tumors (NETs) and neuroendocrine carcinomas (NECs). These are rare malignancies occurring for example in the gastrointestinal tract, islets of the pancreas, lung, adrenal medulla, thyroid C-cells, etc., and is a heterogeneous group of neoplasms with unique tumor biology, natural history, and clinical management issues.
* The annual occurrence of NENs has been increasing in the United States (US) and worldwide. The current incidence in the US is about 6 per 100,000 persons a year and represents 0.46% of all malignancies.
* Most NETs are sporadic, but they can be part of familial cancer syndromes such as multiple endocrine neoplasia type 1 (MEN1), neurofibromatosis type 1 (NF1), or Von Hippel-Lindau (VHL) syndrome. Poorly differentiated NECs are all high-grade carcinomas that resemble small cell carcinoma or large cell NEC of the lung.
* Treatment for localized NETs is surgical resection, however, a variety of therapeutic options are available for patients with advanced NETs. When to apply a given option, what combination therapeutic approach should be used, how long treatment should be continued, and in what subgroup of patients a particular treatment option should be used is unclear and controversial.

Objective:

-To comprehensively and longitudinally evaluate the natural history of participants with NENs and allow sample acquisition for use in the study of NENs

Eligibility:

* Participants with confirmed or suspected NENs including ACC
* Age >=18 years old

Design:

* This protocol is a bio-specimen collection and natural history protocol in which samples will be collected from participants with NENs (from well-differentiated to poorly differentiated neuroendocrine neoplasm).
* An accrual ceiling of 300 participants is planned over an accrual period of 10 years.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age >= 18 years old
* The ability of the participant to understand and the willingness to sign a written consent document.
* Participants with the documentation of:

  * histological or cytological confirmation of NENs or adrenocortical cancer

OR

--biochemical evidence of neuroendocrine tumor (serum/urinary) based on elevated levels of chromogranin A, pancreatic polypeptide, neuron-specific enolase, vasoactive intestinal polypeptide, serotonin (urinary 5-hydroxyindoleacetic acid (5-HIAA)), gastrin, somatostatin, catecholamines, metanephrines, calcitonin, fasting insulin, Cpeptide (proinsulin), glucagon, anterior pituitary hormones

OR

--Suspicion of NEN (from any site/origin) on axial imaging (computed tomography (CT)/ magnetic resonance imaging (MRI) / fluorodeoxyglucose (FDG) positron emission tomography (PET) / 68Ga-Dotatate scan

OR

--a germline genetic variant that predisposes to NETs including ACC.

EXCLUSION CRITERIA:

None

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary clinical
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-04-25 (Actual); Primary Completion 2032-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
natural history of neuroendocrine neoplasms including ACC | ongoing
  To comprehensively and longitudinally evaluate the natural history of participants with NENs and allow sample acquisition for use in the study of NENs

CONTACTS AND LOCATIONS:
Overall Officials: Jaydira Del Rivero, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.@@@@@@In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.@@@@@@Genomic data will be available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.@@@@@@Genomic data will be made available via dbGaP through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000491-C.html